CLINICAL TRIAL: NCT06997445
Title: Additive Effects of Jacobson's Progressive Muscle Relaxation Technique With Aerobic Exercise on Cardiopulmonary Parameters and Quality of Life in Stage 1 Hypertensive Individuals
Brief Title: Jacobson's Progressive Muscle Relaxation Technique With Aerobic Exercise on Cardiopulmonary Parameters and Quality of Life in Stage 1 Hypertensive Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUI/CTR/2024/71
Record Dates: First submitted 2025-05-14; First posted 2025-05-30 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Hypertension
Keywords: aerobic exercise; quality of life; hypertension; Muscle Relaxation
MeSH Terms: conditions — Hypertension | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional group (Active Comparator): Patients in interventional group will receive Jacobson's progressive muscle relaxation technique for 15 minutes and aerobic exercise for 30 minutes.
  For Jacobson's progressive muscle relaxation technique first patient is asked to clench each fist separately, fee the tension, release the fist and relax. Then bend each arm separately, feel the tension and then release the arm. Then straighten the arm separately, feel the tension and then relax. Then wrinkle the forehead, feel the tension and then release the eyebrows relax. Then close the eyes and screw the muscles around the eyes and then release. Then tense the jaw by biting the teeth together and relax. Then press the tongue hard and flat against roof of mouth, feel the tension and then relax. Then push the head back and then bring head back to position. Then bring the head down and then relax. Then shrug the shoulders and relax. Then take a deep breath, hold and then relax. Then tense the stomach muscle and then release. Then arch
  Interventions: Other: Interventional group: Jacobson's progressive muscle relaxation technique with aerobic exercise
- Control group (Other): The control group will receive only aerobic exercise for 45 minutes. Aerobic exercise will include warm uo exercises for 5 minutes, brisk walking on treadmill for 25 minutes which include warm up period for 10 minutes then 14 minutes brisk walk and cool down period included 1 minute walk, stepper for 5 minutes, static cycling for 5 minutes and cool down for 5 minutes.
  Total 4 weeks protocol. Before and after 4 weeks, pre and post intervention values will be taken.
  A total of 20 sessions five days per week for 4 weeks will be provided supervised by physiotherapist
  Interventions: Other: Aerobic Exercise

INTERVENTIONS:
Other: Interventional group: Jacobson's progressive muscle relaxation technique with aerobic exercise — Jacobaon's progressive muscle relaxation technique for 15 minutes Total duration: 45 minutes
  Arms: Interventional group
Other: Aerobic Exercise — Participants in this group will only be provided aerobic exercise for 4 weeks supervised by physiotherapist.
  Aerobic Exercise include the following:
  * Warm up exercises for 5 minutes.
  * Brisk walking on treadmill for 25 minutes which include warm up period for 10 minutes then 14 minutes brisk walk and cool down period included 1 minute walk.
  * Stepper for 5 minutes.
  * Static cycling for 5 minutes.
  * Cool down for 5 minutes.
  Week 03 and Week 04:
  Frequency: 5 days per week Intensity: 60-80% Target heart rate Time: 45 minutes
  Week 01 and Week 02:
  Frequency: 5 days per week Intensity: 50-60 % Target heart rate Time: 45 minutes
  Arms: Control group

SUMMARY:
The study is a randomized controlled trial. The purpose of study is to compare the additive effects of Jacobson's progressive muscle relaxation technique with aerobic exercise versus aerobic exercise on cardiopulmonary parameters including systolic and diastolic blood pressure, heart rate, respiratory rate, rate pressure product and quality of life in stage 1 hypertensive individuals.

DETAILED DESCRIPTION:
The study will consist of referred stage 1 hypertensive patients by medical specialist/cardiologist.

Participants will be screened through PAR-Q and IPAQ Questionnaire. Cardiac monitor will be used for assessing the cardiopulmonary parameters. SF-36 Questionnaire will be used for assessing the quality of life. Informed written consent will be taken after which participants will be recruited into two groups.

Control group will be provided aerobic exercise while interventional group will be provided Jacobson's progressive muscle relaxation technique with aerobic exercise.

Outcome measures assessment will be done at pre-session, at 2 weeks and after 4 weeks post-intervention

ELIGIBILITY:
Inclusion Criteria:

* Adults: aged (18-45 years)
* Gender: both male and female
* Patients diagnosed with stage 1 hypertension (130-139 / 80-89 mmHg according to AHA/ACC 2017 guidelines
* Mild to moderate physical activity level on IPAQ Questionnaire
* Individuals who are able to understand and follow the instructions for exercise

Exclusion Criteria:

* Unstable angina, MI, heart failure, advanced CAD patients
* Severe neurological, musculoskeletal, or gynaecological conditions which limit participation in study
* Recent history of fracture
* Morbidly obese (BMI > 40.0 kg / m2)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2024-08-02 (Actual); Primary Completion 2025-06-05 (Actual); Study Completion 2025-06-05 (Actual)

PRIMARY OUTCOMES:
Systolic and diastolic blood pressure | 04 Weeks
  Evaluation will be done using cardiac monitor for blood pressure.
Heart rate | 04 Weeks
  It will be measured through pulse oximeter.
Respiratory rate | 04 Weeks
  It will be measured by counting the number of breaths a person takes per minute
Rate pressure product | 04 Weeks
  It will be calculated by multiplying heart rate with systolic blood pressure

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University College of Physical Therapy, Islamabad, 44000, Islamabad, Pakistan